CLINICAL TRIAL: NCT00949221
Title: Evaluation of Long-term Efficacy of 2 Strategies of Real Time Continuous Glucose Monitoring, Compared to Self BG-monitoring in Children and Adolescent With Type 1 Diabetes: a Randomized, Multicenter, Open Trial
Brief Title: Study of Insulin Therapy Augmented by Real Time Sensor IN Type 1 Children and Adolescents (START-IN!)
Acronym: START-IN
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P070152; 2007-A01330-53 (Other: IDRCB)
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2023-02-06 (Actual); Status verified 2012-07

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Paediatric; Real Time Continuous Glucose Monitoring; Glycemic control; Therapeutic education
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Other): monitor Paradigm 754 VEO, MINILINK Real Time, Medtronic, CE: Continuous glucose monitoring for 3 months, then conventional blood glucose self-monitoring for 9 months
  Interventions: Device: monitor Paradigm 754 VEO, MINILINK Real Time, Medtronic, CE
- Group 2 (Other): monitor Paradigm 754 VEO, MINILINK Real Time, Medtronic, CE: Intensive strategy using continuous glucose monitoring for 12 months
  Interventions: Device: monitor Paradigm 754 VEO, MINILINK Real Time, Medtronic, CE
- Group 3 (Other): monitor Paradigm 754 VEO, MINILINK Real Time, Medtronic, CE: Intermediate strategy using continuous glucose monitoring for 3 months, then discontinuous use of the device for 9 months (approximately 40% of the time, alternating with conventional blood glucose self-monitoring).
  Interventions: Device: monitor Paradigm 754 VEO, MINILINK Real Time, Medtronic, CE

INTERVENTIONS:
Device: monitor Paradigm 754 VEO, MINILINK Real Time, Medtronic, CE — * group 1: continuous glucose monitoring for 3 months, then conventional blood glucose self-monitoring for 9 months;
  * group 2: intensive strategy using continuous glucose monitoring for 12 months;
  * group 3: intermediate strategy using continuous glucose monitoring for 3 months, then discontinuous use of the device for 9 months (approximately 40% of the time, alternating with conventional blood glucose self-monitoring).

SUMMARY:
Glycemic control in children and adolescent with type 1 diabetes remains inadequate, exposing them to the risk of vascular complications in adulthood.

One of the limiting factors is the daily number of self measurements of blood glucose required to optimize intensive insulin therapy.

Real Time Continuous Glucose Monitoring augmented by alarms (RT CGM) is a recent innovation. A randomized clinical study has shown its efficacy at short term (3 months). However, optimal clinical use of these devices requires rigorous assessment of their effectiveness on glycemic control, tolerance and acceptability in medium and long term.

Primary objective: To assess the long-term effectiveness of two strategies of use of RT CGM (continuous or discontinuous) on glycemic control compared to conventional blood glucose self-monitoring (SMBG).

Population: Children and adolescents with type 1 diabetes with inadequate glycemic control despite intensive insulin therapy.

DETAILED DESCRIPTION:
Despite the development of intensive insulin therapy, glycemic control defined by glycated haemoglobin (HbA1c) < 7,5% remains inadequate in pediatric patients with type 1 diabetes.

Improvement of the metabolic control is limited by the daily number of self measurements of blood glucose required to adjust closely insulin therapy

Improving glycemic control is particularly important in type 1 children and adolescent, whose risk of vascular complications in adulthood is high, due to the duration of the disease and whose adherence to current strategies of blood glucose self-monitoring is limited.

Real Time Continuous Glucose Monitoring augmented by alarms (RT CGM) is a recent innovation. A randomized clinical study has shown improvement of HbA1c (≈ 1%) without increasing frequency of hypoglycaemia after continuous use for 3 months. Optimal clinical use of these new devices requires rigorous assessment of their effectiveness on glycemic control, tolerance and acceptability at medium and long term.

Primary objective: To assess the long-term effectiveness of two strategies of use of RT CGM on glycemic control compared to conventional blood glucose self-monitoring.

Secondary objectives: overall comparison of 2 strategies of continuous use of RT CGM vs conventional SMBG on HbA1c ; to evaluate their effectiveness on others parameters of glycemic control (hypoglycaemias, ketoacidosis, glycemic variability); to evaluate impact on glycemic control of different factors including percentage of effective time of wearing the sensor; to evaluate : skin tolerance, acceptability of the device; quality of life and satisfaction to the use of the device; and medico-economic impact of the use of the device.

Population: Type 1 diabetes children and adolescent with inadequate metabolic control despite intensive insulin therapy, randomized in 3 groups. After a period of 3 months of continuous measurement for all of them, the two strategies will be an intensive glucose monitoring by continuous measurement for 9 months (a total of 12 months) and an intermediate consisting of discontinuous measurement (40% of the time for 9 months), compared to conventional blood glucose self-monitoring.

The reduction in HbA1c of at least 0,6% requires 50 patients per group, and a total of 150 children.

Primary endpoint: change in the rate of HbA1c.

Secondary endpoints: frequency of acute metabolic events, non-severe or symptomatic hypoglycaemia; measure of glycemic variability; skin tolerance; number of sensor used and percentage of effective time of use of the device; satisfaction of the patients; quality of life and diabetes-related quality of life; choice of the patient (continuing or not to use the device) at the end of the study; medico-economic evaluation.

Benefits expected with this clinical trial: improvement of glycemic control and quality of life in children and adolescents with type 1 diabetes. Furthermore, study results would permit to defined optimal strategy of using RT CGM in paediatric population.

ELIGIBILITY:
Inclusion Criteria:

* Age between 2 years and 17 years 11 months.
* Onset of type 1 diabetes ≥ 1 year.
* Centralized HPLC HbA1c ≥ 7.5% and < 11%.
* Intensive insulin therapy either by multiple daily injections ≥ 3 / day (rapid insulin analogue before 3 meal and 1 to 2 injections of basal insulin) or by continuous subcutaneous insulin infusion (pump).
* Followed in the centre for ≥ 3 months.
* Blood glucose self-monitoring ≥ 2/day.
* No significant change of regimen insulin therapy for at least 3 months.
* Patient receiving medical health insurance.
* Patient who has given his consent

Exclusion Criteria:

* Non type 1 diabetes(type 2 diabetes or diabetes whose evolution suggest other origin).
* Association with another pathology which, in the discretion of the investigator, could affect the monitoring or be disturbed by the participation in the study.
* Association with chronic treatment (steroids, growth hormone…) or chronic disease, including hypothyroidism and celiac disease, non stabilized for 3 months.
* Association with severe skin disease.
* Deafness, hearing or visual defect.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2009-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Comparison of the effect of 2 strategies of real time continuous glucose monitoring vs conventional SMBG on glycated haemoglobin = HbA1c measured at inclusion, 3, 6, 9, 12 months | 1 year

SECONDARY OUTCOMES:
HbA1c and associated factors with HbA1c changes, others parameters of glycemic control, tolerance, acceptability, quality of life, satisfaction after use of real time continuous glucose monitoring in 150 pediatric patients | 3 months
Frequency of acute metabolic events (severe hypoglycaemia or ketoacidosis) | 1 year
Frequency of non-severe or symptomatic hypoglycaemia | 1 year
Average blood glucose and glycemic variability | 1 year
Tolerance of using the device of continuous glucose monitoring (skin tolerance) | 1 year
Acceptability of the device (percentage of time of use) | 1 year
General and diabetes-related Quality of life | 1 year
Satisfaction to use the device | 1 year
Medico-economic evaluation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Tubiana, PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Robert Debré, Paris, France

REFERENCES:
- [Result] Guilmin-Crepon S, Carel JC, Schroedt J, Scornet E, Alberti C, Tubiana-Rufi N. How Should We Assess Glycemic Variability in Type 1 Diabetes? Contribution of Principal Component Analysis for Interstitial Glucose Indices in 142 Children. Diabetes Technol Ther. 2018 Jun;20(6):440-447. doi: 10.1089/dia.2017.0404. PMID 29923773
- [Result] Guilmin-Crepon S, Carel JC, Schroedt J, Sulmont V, Salmon AS, Le Tallec C, Coutant R, Dalla-Vale F, Stuckens C, Bony-Trifunovic H, Crosnier H, Kurtz F, Kaguelidou F, Le Jeannic A, Durand-Zaleski I, Couque N, Alberti C, Tubiana-Rufi N. Is there an optimal strategy for real-time continuous glucose monitoring in pediatrics? A 12-month French multi-center, prospective, controlled randomized trial (Start-In!). Pediatr Diabetes. 2019 May;20(3):304-313. doi: 10.1111/pedi.12820. Epub 2019 Feb 6. PMID 30663187
- [Result] Le Jeannic A, Maoulida H, Guilmin-Crepon S, Alberti C, Tubiana-Rufi N, Durand-Zaleski I. How to collect non-medical data in a pediatric trial: diaries or interviews. Trials. 2020 Jan 7;21(1):36. doi: 10.1186/s13063-019-3997-9. PMID 31910885